CLINICAL TRIAL: NCT04381598
Title: Efficacy of Stevia Rebaudiana Bertoni on Levels of GCF Glucose and Bio-markers in Diabetic Patients With Periodontitis-A Split Mouth Randomized Controlled Trial.
Brief Title: Stevia Rebaudiana Bertoni on Levels of GCF Glucose and Bio-markers in Diabetics.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: SVS Institute of Dental Sciences (Other)
Responsible Party: Principal Investigator, Dr R Viswa Chandra, Principal Investigator, SVS Institute of Dental Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: SVSIDS/perio/3/2019
Record Dates: First submitted 2020-04-29; First posted 2020-05-11 (Actual); Last update posted 2020-05-11 (Actual); Status verified 2020-05

CONDITIONS: Periodontitis
Keywords: Biomarkers; Gingival crevicular fluid; Glucose; Diabetes
MeSH Terms: conditions — Periodontitis; Diabetes Mellitus | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: one group of subjects receives intervention where as other group of subjects receive placebo.
Who Masked: Participant, Investigator
Masking Description: Both stevia gel and placebo syringes are masked from participants and investigators.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- stevia rebaudiana bertoni (Experimental): Randomly in all subjects one quadrant will be allotted as test site for placing stevia gel in the gingival sulcus having probing depth ≥ 5mm after performing thorough scaling and root planing.
  Interventions: Drug: stevia rebaudiana bertoni
- placebo (Placebo Comparator): Other quadrant will be allotted as a control site for placing placebo in the gingival sulcus having PD≥ 5mm after performing thorough scaling and root planing.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: stevia rebaudiana bertoni — Stevia has an anti-plaque effect because of its ability in decreasing the formation of bacterial insoluble polymers.It significantly decreases the production of TNF-R and IL-1a and slightly decreases the production of NO in stimulated cells with LPS and THP-1 showing its anti-inflammatory properties.These characteristics in combination with anti-diabetic properties could results in the effective treatment of periodontal diseases.
  Other Names: sweet tulasi
  Arms: stevia rebaudiana bertoni
Other: placebo — A placebo without the active drug will be placed in the control sites.
  Other Names: Control group
  Arms: placebo

SUMMARY:
With the increase in the incidence of diabetes and obesity, among other artificial sweeteners the need of natural non-caloric sweetener with acceptable taste and without any adverse effects is demanding.So,the use of stevia presents beneficial effects to general and oral health and its properties could result potentially effective in the treatment of periodontal diseases.

DETAILED DESCRIPTION:
Stevia is considered as a novel molecule, because it is 100% natural and non caloric sweetener, with more sweetness than sucrose, without any adverse effects. It also demonstrates multiple benefits like anti-plaque effect, anti-diabetic effect, anti-periodontophatics properties, anti-hypertensive properties, anti-cariogenic properties etc. There are many studies conducted on stevia in humans, which justifies my study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects that will be included in the study are in the age group ranging from 20-70 years -with established diabetes and under medication to maintain normal glycemic state i.e;Hb1Ac < 7％.
* Oral findings including the presence of minimum of 16 natural teeth with minimum of 4 nonadjacent sites showing pocket depths≥ 5 mm.

Exclusion Criteria:

Subjects will be excluded from the study if they are using

* any type of mouth-rinses or if they had underwent any periodontal therapy within the 3-months of the study or
* if they were under antibiotics within the 3-months of the study.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-10 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Bio-marker (Ghrelin) levels in Gingival crevicular fluid. | From baseline to 6-months.
  GCF samples can be eluted from the strips by placing them in Eppendrof® tubes that contained 500 micro-litre of buffer and will be stored at -80℃ until analysis was done. The levels of GCF Ghrelin will be evaluated by using commercially available ELISA kit.

SECONDARY OUTCOMES:
Probing depth | From baseline to 6-months.
  Probing depth (PD): Distance from the gingival margin to the bottom of gingival sulcus in mm.

CONTACTS AND LOCATIONS:
Locations (1):
- SVS Institute Of Dental Sciences, Hyderabad, Telangana, India